CLINICAL TRIAL: NCT05477329
Title: EVALUATING THE EFFECT OF A MYOPIA CONTROL SPECTACLE LENS COMPARED TO A SINGLE VISION SPECTACLE LENS AMONG CHILDREN IN ISRAEL
Brief Title: CHILDREN MYOPIA CONTROL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shamir Optical Industry Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MCIS2021
Record Dates: First submitted 2022-07-26; First posted 2022-07-28 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Myopia
Keywords: MYOPIA CONTROL
MeSH Terms: conditions — Myopia | interventions — Lenses

STUDY DESIGN:
Intervention Model Description: This will be a controlled, randomized, double-masked trial. The Test group will wear the myopia control spectacle lens and the Control group will wear the single vision spectacle lens.
Who Masked: Participant, Care Provider, Investigator
Masking Description: This will be a controlled, randomized, double-masked trial. The Test group will wear the myopia control spectacle lens and the Control group will wear the single vision spectacle lens.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myopia control design spectacle lens (Experimental): Test lenses
  Interventions: Device: Lenses
- Single Vision design spectacle lens (Other): Control lenses
  Interventions: Device: Lenses

INTERVENTIONS:
Device: Lenses — The test lens is manufactured in a standard FreeForm technology (exactly like a standard progressive addition lens which is similar in terms of the graduall power profile induced in both lens). It does not demand any special manufacturing processes.

SUMMARY:
The purpose of this trial is evaluating the clinical effect of a myopia control spectacle lens compared to a single vision spectacle lens in slowing down the progression of myopia in children living in Israel.

DETAILED DESCRIPTION:
TRIAL PLAN

Screening visit (VISIT 1)

* Enrollment criteria verification
* Signing informed consent
* Baseline documentation of medical history, parental and siblings myopia, indoor and outdoor activities profile and socioeconomic profile
* Lensmeter measurements of participants spectacles
* Performing baseline measurements including best corrected VA, objective & subjective refraction under cycloplegia, PR under cycloplegia*, slit lamp examination, functional tests: cover test, titmus test, worth four dot test, axial length** and pupil size measurements
* Frame selection and frame measurements
* Lens order completion and sending to manufacturing

Randomization Procedures (following VISIT 1) Randomization procedures should be performed by the trial coordinator following visit 1. The participant will then be allocated to the test or control group.

Manufacturing Procedures (following VISIT 1) The manufacturing technician will take care of the manufacturing processes according to the lens type (test or control) and the mounting on the frame. The test spectacles will then be sent to the site for delivery.

Delivery visit (VISIT 2) performed ~10 days after screening visit

* Trial spectacles delivery
* Subjective questionnaire while wearing the trial spectacles
* Best corrected far and near VA (with the trial spectacles)
* Confrontation visual field test with the trial spectacles
* Giving instructions about wearing the trial spectacles
* Documenting adverse events if relevant

Follow-up visit performed 6 months (±1 week) after the previous visit (VISITS 3,4,5,6)

* Documentation of any change medical history since last visit
* Subjective questionnaire regarding the wearing period with the trial spectacles (feedback performing follow-up measurements including best corrected far and near VA, objective & subjective refraction under cycloplegia, PR under cycloplegia*, slit lamp examination, functional tests: cover test, titmus test, worth four dot test, axial length and pupil size measurements
* If the subjective refraction will find a SE (Sphere Equivalent) change from last refraction of at least -0.50D, a new lens order should be made for new lenses, and a delivery visit should be set in order to deliver the new test spectacles. The procedures mentioned above in the delivery visit (visit 2) should then be performed.
* Documenting adverse events if relevant

Additional unscheduled visits

* May be scheduled as needed if special needs occur
* Procedures will be defined by the investigator
* Documenting adverse events if relevant

Total duration of trial per patient: 24 months.

ETHICAL ISSUES

This trial will be conducted according to the applicable local regulations and the GCP. All essential documents will be reviewed and approved by the ethics committee prior to the beginning of the trial. Any amendments of these documents will be reviewed and approved by the ethics committee prior to implantation in the trial.

Informed Consent The investigator will give the participant and their parent/legal guardian a full explanation about the trial and will answer all their question regarding participating in the trial.

The investigator will explain that the participant will be able to withdraw from the trial at any stage for any reason.

The participants parent/legal guardian will sign the informed consent form and will receive a signed copy of it.

Data confidentiality All identification details about the participants in the trial will be held by the investigator in a secured log file kept at the trial site.

Access to the identification details will not be allowed to any unauthorized party and will not be disclosed in any report/document relating to the trial.

Terminating the participation in the trial

These are the cases in which an early termination of the participation in the trial may occur:

1. Should the myopia progression of the participant will be more than 1.00 D after 1 year or other significant refractive changes (such as more than 0.5[D] cylinder) - the investigator will recommend the participant to discontinue the participation in the trial and to consider using other myopia control treatments such as low dose Atropine drops.
2. Should the far/near VA with the trial spectacles will be less than the best corrected VA of the participant, the investigator will consider recommending the participant to discontinue the participation in the trial.

RISK EVALUATION/ ADVERSE EVENTS

The optical design of the test lens, with the gradual positive peripheral power, induce a certain amount of aberrations in the peripheral areas of the lens. These aberrations were designed such that a good level of compliance will be achieved so that the participant will be able to wear the lens.

Adverse events are unlikely to occur, yet it should be mentioned that a participant should not wear this lens in case of one/more of the following exist:

* Feeling significant amount of discomfort while wearing the lens such that the safety of the participant might be at risk.
* Vestibular disorders The participants in the trial will be free to contact the investigator at any time during the wearing period in order to report any unexpected events that might occur. The investigator will decide based on the report whether the child should be excluded from continuing the trial.

Furthermore, it should be noted that a parallel clinical trial is being conducted these days in AIER hospital in China, managed and supervised by Brien Holden Vision Institution (Australia). The trial is similar to our trial, with the same trial product, on a group of 140 participants with the same enrollment criteria, including similar trial procedures and trial plan. The trial started at November 2020, and as for now most of the participants has worn the test spectacles for a few months with no adverse events reported.

DATA MANAGEMENT

Database An electronic data base will be held and maintained, into which all the source data will be electronically transferred from the measuring devices, or if not possible, will be typed in and source data (printouts or location of data) will be kept in the participants file. At any case, all source data (printouts or location of data) should be kept in the participants file.

The electronic data base will be backed up on a daily basis

Access to data:

The investigator will be able to allow access to data to the Sponsor (without identification data) as per request.

The investigator will be able to allow access to data to the Monitoring staff according to the monitoring plan that will be defined.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent form signed and fully comprehended by the parent/legal representative of the participant
* Age from 6 to 12 years old
* Both male and female
* Spherical Equivalent refractive error (cycloplegic objective) of -0.50D to -5.00D
* Astigmatism not higher than -1.50D
* Corrected Visual Acuity of not less than 6/7.5 or 20/25
* Willing to wear the trial spectacles for the defined period according the protocol plan

Exclusion Criteria:

* Current participation in another clinical trial
* Any general health or ocular health pathology that could affect the treatment
* Allergy or intolerance to cycloplegic eye drops (name should be stated here)
* Strabismus
* Amblyopia
* History of ocular injury or ocular surgery
* Previously been treated with any myopia control treatments (Orthokeratology, myopia control spectacle/contact lenses, multifocal lenses, bifocal lenses, atropine)

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 136 (Actual)
Dates: Start 2021-06-20 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Refractive error | 3 seconds
  Objective cycloplegic refractive error (Sphere equivalent)

SECONDARY OUTCOMES:
Axial length | 3 seconds

CONTACTS AND LOCATIONS:
Locations (1):
- "Maor" Institute Clinic, Rishon LeZiyyon, Israel